CLINICAL TRIAL: NCT04009863
Title: A Randomized, Open-label, Parallel-group Study to Determine the Efficacy of Sequential High-intensity Focused Ultrasound (HIFU) Ablation Versus Fixed-dose Radioiodine-131 Therapy in Moderate-sized Non-toxic Multinodular Goiter
Brief Title: HIFU Ablation vs Fixed-dose RAI-131 Therapy in Moderate-sized Non-toxic MNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UW 19-016
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Non Toxic Multinodular Goiter; High Intensity Focused Ultrasound; RAI

STUDY DESIGN:
Intervention Model Description: group 1 is for HIFU treatment, group 2 is for RAI treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFU on NMNG (Active Comparator): The patients with non-toxic multinodular goiter are assigned to have high intensity focused ultrasound treatment.
  Interventions: Device: Echopulse
- RAI on NMNG (Active Comparator): The patients with non-toxic multinodular goiter are assigned to have radioactive iodine (i131) treatment.
  Interventions: Radiation: Radioactive iodine (Radioidine i131)

INTERVENTIONS:
Device: Echopulse — Echopulse is a real-time US-guided High-intensity focused ultrasound (HIFU) system, the HIFU session is a noninvasive procedure that involves application of a focused high-energy ultrasound beam for thermal tissue ablation inside the targeted zone, with minimal effect on the surrounding tissue
  Other Names: High Intensity Focused Ultrasound (HIFU)
  Arms: HIFU on NMNG
Radiation: Radioactive iodine (Radioidine i131) — Radioactive iodine (RAI) is a radioactive form of iodine that for ablation in thyroid disease (i.e. Graves' disease or few thyroid cancer)
  Arms: RAI on NMNG

SUMMARY:
After obtaining informed consent, eligible subjects will be assigned randomly into either High intensity focused ultrasound group (HIFU) or Radioactive iodine (131I) therapy group (RAIT). After treatment, they will be followed up for 4 visits (1-month, 3-month, 6- month, 12-month of post treatment). At each visit, they will have physical examination, regular blood test and questionnaire to evaluate their quality of life. The collected data will be used to compare the effectiveness between HIFU and RAIT for non-toxic multi-nodular goiter (NMNG). The primary purepose is to find out the best non-invasive way in treating NMNG.

For HIFU, you may experience:

1. Mild bruising and redness at the site of treatment
2. Edema of the skin tissue
3. Pain/discomfort during the procedure
4. Skin burns but rare (<1%)
5. Vocal cord paresis on the side of the treated lobe but rare (<1%)
6. Unintentional damage to the surrounding tissue (outside the planned treatment area).

For RAIT, you may experience neck tenderness or sore throat in the following few days as developing moderate inflammation in the thyroid and producing discomfort in the neck or throat area. Your symptoms may turn worse for first few week, but will improve over weeks.

DETAILED DESCRIPTION:
Non-toxic multinodular goiter (NMNG) is a condition referred to as a nodular enlargement of the thyroid gland due to the presence of two or more nodules without clinical hyper- or hypothyroidism. It is undoubtedly one of the most common thyroid disorders worldwide and it is estimated that more than 5% of the female population have a clinically-palpable NMNG (1,2).

Although the majority of NMNGs do not cause symptoms and therefore, do not require any intervention other than simple surveillance, some can cause local pressure symptoms and cosmetic concerns over time (1-3).

For NMNGs that cause symptoms, the most widely-accepted treatment has been surgical resection either in the form of a hemithyroidectomy or total thyroidectomy. Despite being safe when done in experienced hands, surgery is associated with complications such as recurrent laryngeal nerve injury and hypoparathyroidism, both of which can be permanent. In addition, a general anesthesia is almost inevitably required when surgery is performed. As a result, non-surgical thermal ablation techniques have been increasingly recognized as an alternative treatment in symptomatic NMNG (4). These ablation techniques utilize thermal energy to cause shrinkage of adenomatous nodules and thereby, relieve symptoms. Types of ablation include radiofrequency, laser and microwave ablations and more recently, high intensity focused ultrasound (HIFU). Regardless of which ablation technique, they have all been shown to not only induce significant nodule shrinkage but also alleviate symptoms (4-6). Radioactive iodine (131I) therapy (RAIT) is another promising non-surgical alterative which is recommended in patients who refuse or have contraindications for surgery. Despite being a less recognized treatment in both Asia and North America, this treatment has increasingly been adopted. In some European countries such as Denmark and Netherlands, it has replaced surgery as the treatment of choice in moderately-sized NMNG as recommended in recently-published clinical practice guidelines (1,7,8). However, RAIT has limitations. For example, it is less applicable in very large-sized NMNG (>100 mL) because large goiters tend to have a lower radioiodine uptake leading to suboptimal shrinkage. Also considerable inconsistency in goiter shrinkage has been reported (7). With our population getting older and the general public placing a greater emphasis on preserving organ function and lessinvasive treatments, non-surgical treatment alternatives will have an increasing role in the future treatment of NMNG. To our knowledge, it remains unknown whether one particular treatment modality is superior over the other modality because there has not been any direct comparison between the two modalities. Only one previous study compared treatment efficacy between laser ablation and RAIT. However, it mainly focused on the treatment of toxic thyroid nodules (9). To enhance treatment efficacy, a recent study reported promising results of combining the effect of thermal ablation and RAIT (10).

ELIGIBILITY:
Inclusion Criteria:

* Have a moderate-sized NMNG. The dimension of the largest nodule cannot exceed 50mm in diameter. Also on USG volumetry, the total combined volume of the three largest nodules (i.e. the largest nodule volume + second largest nodule volume + third largest nodule volume) or in short, TNV cannot exceed 80 mL or cm^3.
* The NMNG has to benign. Each nodule within the goiter will be carefully evaluated on USG by an experienced clinician to look for suspicious features for malignancy. Suspicious-looking nodules will be biopsied by USG-guided FNAC. Only nodules with Bethesda II on FNAC will be considered benign.
* Aged between 18 and 70 years old at the time of informed consent.
* Have genuine cosmetic and/or pressure symptoms.
* Have to have normal serum free T4 (FT4) and thyroid-stimulating hormone (TSH) levels.

Exclusion Criteria:

* Have a non-toxic diffuse goiter or a NMNG with the largest nodule < 20mm in diameter.
* Prefer or have a clear indication for thyroidectomy (such as rapidly growing, compressive goiter or suspected or documented thyroid malignancy).
* Have a pre-existing vocal cord palsy.
* Unable to tolerate even slight neck extension during HIFU ablation.
* Pregnant, lactating women or women wishing to become pregnant within 6 months.
* Previous thyroid surgery or neck irradiation.
* Family history of non-medullary thyroid carcinoma.
* Have any medical conditions that would make them too ill to undergo treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The absolute change in Thyroid nodule volume (TNV) after sequential HIFU treatment and a fixed-dose (370MBq) RAIT after 12 months. | 12 months
  To compare the absolute change in Thyroid nodule volume (in cm^3) after sequential HIFU treatment and a fixed-dose (370MBq) RAIT after 12 months.

SECONDARY OUTCOMES:
Change in total thyroid volume (TTV) (in cm^3) | 12 months
  To compare the absolute change in TTV between HIFU and RAIT groups
Change in the largest/dominant nodule dimensions | 12 months
  To compare the change in the largest/dominant nodule dimensions (in cm) between HIFU and RAIT groups
Incidence of treatment-related morbidities after HIFU/RAIT | 12 months
  To compare incidence of treatment-related morbidities and hypothyroidism between HIFU and RAIT groups
Change in World Health Organization goiter grade | 12 months
  To compare WHO goiter grade over time between HIFU and RAIT groups
Change in symptom improvement score | 12 months
  To compare symptom improvement score (0-10) over time between HIFU and RAIT groups
Change in pressure symptom score | 12 months
  To assess the changes in pressure symptom score (by Visual Analogue Scale, VAS, scoring from 0-10, 0 is for no pressure and 10 is for the maximum pressure feeling as subjects' view) over time between the HIFU and RAIT groups.
Change in quality of life | 12 months
  To assess the changes in quality of life (QOL) using by "12-Item Short Form Survey (SF-12) (VERSION 2.0)" between the two treatment groups. SF-12 is scoring 70 in total, the higher score represent higher quality of life.
Change in patient satisfaction | 12 months
  To assess the changes in patient satisfaction (by Visual Analogue Scale, VAS, scoring from 0-10, 10 is for the maximum score representing well satisfaction) between the two treatment groups
Compare the costs (in dollars) | 12 months
  To compare the direct and indirect costs between HIFU and RAIT (in dollars)

CONTACTS AND LOCATIONS:
Overall Officials: Hung Hin Brian Lang, MBBS(Hons), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Gharib H, Papini E, Garber JR, Duick DS, Harrell RM, Hegedus L, Paschke R, Valcavi R, Vitti P; AACE/ACE/AME Task Force on Thyroid Nodules. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS, AMERICAN COLLEGE OF ENDOCRINOLOGY, AND ASSOCIAZIONE MEDICI ENDOCRINOLOGI MEDICAL GUIDELINES FOR CLINICAL PRACTICE FOR THE DIAGNOSIS AND MANAGEMENT OF THYROID NODULES--2016 UPDATE. Endocr Pract. 2016 May;22(5):622-39. doi: 10.4158/EP161208.GL. PMID 27167915
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Durante C, Costante G, Lucisano G, Bruno R, Meringolo D, Paciaroni A, Puxeddu E, Torlontano M, Tumino S, Attard M, Lamartina L, Nicolucci A, Filetti S. The natural history of benign thyroid nodules. JAMA. 2015 Mar 3;313(9):926-35. doi: 10.1001/jama.2015.0956. PMID 25734734
- [Background] Gharib H, Hegedus L, Pacella CM, Baek JH, Papini E. Clinical review: Nonsurgical, image-guided, minimally invasive therapy for thyroid nodules. J Clin Endocrinol Metab. 2013 Oct;98(10):3949-57. doi: 10.1210/jc.2013-1806. Epub 2013 Aug 16. PMID 23956350
- [Background] Sung JY, Baek JH, Kim KS, Lee D, Yoo H, Kim JK, Park SH. Single-session treatment of benign cystic thyroid nodules with ethanol versus radiofrequency ablation: a prospective randomized study. Radiology. 2013 Oct;269(1):293-300. doi: 10.1148/radiol.13122134. Epub 2013 Apr 24. PMID 23616630
- [Background] Lang BH, Woo YC, Wong CKH. High-Intensity Focused Ultrasound for Treatment of Symptomatic Benign Thyroid Nodules: A Prospective Study. Radiology. 2017 Sep;284(3):897-906. doi: 10.1148/radiol.2017161640. Epub 2017 Apr 18. PMID 28419814
- [Background] Bonnema SJ, Hegedus L. Radioiodine therapy in benign thyroid diseases: effects, side effects, and factors affecting therapeutic outcome. Endocr Rev. 2012 Dec;33(6):920-80. doi: 10.1210/er.2012-1030. Epub 2012 Sep 7. PMID 22961916
- [Background] Paschke R, Hegedus L, Alexander E, Valcavi R, Papini E, Gharib H. Thyroid nodule guidelines: agreement, disagreement and need for future research. Nat Rev Endocrinol. 2011 Jun;7(6):354-61. doi: 10.1038/nrendo.2011.1. Epub 2011 Mar 1. PMID 21364517
- [Background] Dossing H, Bennedbaek FN, Bonnema SJ, Grupe P, Hegedus L. Randomized prospective study comparing a single radioiodine dose and a single laser therapy session in autonomously functioning thyroid nodules. Eur J Endocrinol. 2007 Jul;157(1):95-100. doi: 10.1530/EJE-07-0094. PMID 17609407
- [Background] Mader A, Mader OM, Groner D, Korkusuz Y, Ahmad S, Grunwald F, Kranert WT, Happel C. Minimally invasive local ablative therapies in combination with radioiodine therapy in benign thyroid disease: preparation, feasibility and efficiency - preliminary results. Int J Hyperthermia. 2017 Dec;33(8):895-904. doi: 10.1080/02656736.2017.1320813. Epub 2017 May 5. PMID 28540810
- [Background] Lang BHH, Woo YC, Chiu KW. Sequential high intensity focused ultrasound (HIFU) ablation in the treatment of benign multinodular goitre: an observational retrospective study. Eur Radiol. 2018 Aug;28(8):3237-3244. doi: 10.1007/s00330-018-5333-2. Epub 2018 Mar 19. PMID 29556769
- [Background] Lang BH, Woo YC, Chiu KW. Single-Session High-Intensity Focused Ultrasound Treatment in Large-Sized Benign Thyroid Nodules. Thyroid. 2017 May;27(5):714-721. doi: 10.1089/thy.2016.0664. Epub 2017 Mar 22. PMID 28326895
- [Background] Eng OS, Potdevin L, Davidov T, Lu SE, Chen C, Trooskin SZ. Does nodule size predict compressive symptoms in patients with thyroid nodules? Gland Surg. 2014 Nov;3(4):232-6. doi: 10.3978/j.issn.2227-684X.2014.08.03. PMID 25493254
- [Background] Zimmermann M, Saad A, Hess S, Torresani T, Chaouki N. Thyroid ultrasound compared with World Health Organization 1960 and 1994 palpation criteria for determination of goiter prevalence in regions of mild and severe iodine deficiency. Eur J Endocrinol. 2000 Dec;143(6):727-31. doi: 10.1530/eje.0.1430727. PMID 11124854
- [Background] Lang BHH, Woo YC, Chiu KW. Significance of hyperechoic marks observed during high-intensity focused ultrasound (HIFU) ablation of benign thyroid nodules. Eur Radiol. 2018 Jun;28(6):2675-2681. doi: 10.1007/s00330-017-5207-z. Epub 2018 Jan 8. PMID 29313120
- [Background] Wong KP, Lang BH, Ng SH, Cheung CY, Chan CT, Lo CY. A prospective, assessor-blind evaluation of surgeon-performed transcutaneous laryngeal ultrasonography in vocal cord examination before and after thyroidectomy. Surgery. 2013 Dec;154(6):1158-64; discussion 1164-5. doi: 10.1016/j.surg.2013.04.063. Epub 2013 Aug 19. PMID 23969288
- [Background] Royal College of Physicians. Radioiodine in the management of benign thyroid disease: clinical guidelines. Report of a Working Party. London: RCP, 2007. Available from: http://www.thyroiduk.org.uk/tuk/guidelines/Radioiodine%20guidelines%202007.pdf
- [Background] Hospital Authority. 2013. Revisions to List of charges: G.N. 1488 to Gazette No. 12/2013. In Hong Kong Government Printers. Available: http://www.gld.gov.hk/egazette/english/gazette/toc.php [Accessed at 1st February 2018]